CLINICAL TRIAL: NCT04625972
Title: A Phase III Randomized, Double-blind, Placebo-controlled, Multi-center Study in Adults to Determine the Safety and Efficacy of AZD7442, a Combination Product of Two Monoclonal Antibodies (AZD8895 and AZD1061), for Post-exposure Prophylaxis of COVID-19
Brief Title: Phase III Double-blind, Placebo-controlled Study of AZD7442 for Post- Exposure Prophylaxis of COVID-19 in Adults
Acronym: STORM CHASER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D8850C00003; 2020-004719-28 (EudraCT Number)
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: Post exposure COVID-19
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination; tixagevimab; cilgavimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AZD7442 (Experimental): Participants will be randomized in a 2:1 ratio to receive a single dose (× 2 IM injections) of either 300 mg of AZD7442 (n = approximately 750) or saline placebo (n = approximately 375) on Day 1.
  Interventions: Drug: AZD7442
- Placebo (Placebo Comparator): Participants will be randomized in a 2:1 ratio to receive a single dose (× 2 IM injections) of either 300 mg of AZD7442 (n = approximately 750) or saline placebo (n = approximately 375) on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7442 — Single dose (× 2 IM injections) of 300 mg of AZD7442 on Day 1.
  Other Names: A combination of 2 mAbs (AZD8895 and AZD1061)
  Arms: AZD7442
Drug: Placebo — Single dose (× 2 IM injections) of saline placebo on Day 1.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy of AZD7442 for the post-exposure prophylaxis of COVID-19 in Adults.

DETAILED DESCRIPTION:
SARS-CoV-2 is the causative agent of the ongoing COVID-19 pandemic that, as of 29 September 2020, has resulted in a high death toll to date. Unlike the majority of coronaviruses that cause mild disease in humans and animals, SARS-CoV-2 can replicate in the lower respiratory tract to cause acute respiratory distress syndrome and fatal pneumonia. Effective interventions to prevent or treat COVID-19 remain limited in number and clinical experience is limited. Clinical management is limited to supportive care, consequently overwhelming resources of healthcare systems around the world. As a response to the ongoing pandemic, AstraZeneca is developing mAbs to the SARS-CoV-2 S protein. The SARS-CoV-2 spike protein contains the virus's RBD, which enables the virus to bind to receptors on human cells. By targeting this region of the virus's spike protein, antibodies can block the virus's attachment to human cells, and, therefore, is expected to block infection. Amino acid substitutions have been introduced into the antibodies to both extend their half-lives, which should prolong their potential prophylactic benefit, and decrease Fc effector function in order to decrease the potential risk of antibody-dependent enhancement of disease. AZD7442, a combination of 2 of these mAbs (AZD8895 and AZD1061), is being evaluated for administration to prevent and/or treat COVID-19. There is currently one ongoing Phase I study with AZD7442.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of signing the informed consent
2. Adults with potential exposure, within 8 days, to a specific identified individual with laboratory-confirmed SARS-COV-2 infection, symptomatic or asymptomatic
3. Participants must not have had COVID-19 symptoms within 10 days of dosing
4. Negative result from point of care SARS-CoV-2 serology test at screening
5. Contraception used by women of childbearing potential, condom by men
6. Able to understand and comply with study requirements/procedures based on the assessment of the investigator

Exclusion Criteria:

1. History of laboratory-confirmed SARS-CoV-2 infection or SARS-CoV-2 seropositivity at screening.
2. History of infection with severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS).
3. Known history of allergy or reaction to any component of the study drug formulation.
4. Previous hypersensitivity, infusion-related reaction, or severe adverse reaction following administration of a mAb.
5. Any prior receipt of investigational or licensed vaccine or other mAb/biologic indicated for the prevention of SARS-CoV-2 or COVID-19 or expected receipt during the period of study follow up.
6. Clinically significant bleeding disorder or prior history of significant bleeding or bruising following IM injections or venipuncture.
7. Any other significant disease, disorder, or finding that, in the judgement of the investigator, may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study, or impair interpretation of the study data.
8. Receipt of any IMP in the preceding 90 days or expected receipt of IMP during the period of study follow-up, or concurrent participation in another interventional study.
9. Currently pregnant or breast feeding.
10. Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 30 days prior to randomization.
11. Employees of the Sponsor involved in planning, executing, supervising, or reviewing the AZD7442 program, clinical study site staff, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
12. In nations, states, or other jurisdictions that for legal or ethical reasons bar the enrollment of participants who lack capacity to provide their own informed consent, such subjects are excluded.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1131 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Levin, MD, Principal Investigator — AstraZeneca
Locations (50):
- United States (45):
  - Research Site, Guntersville, Alabama
  - Research Site, Tempe, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Corona, California
  - Research Site, Garden Grove, California
  - Research Site, Huntington Beach, California
  - Research Site, Huntington Park, California
  - Research Site, Modesto, California
  - Research Site, Coral Gables, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Mt. Dora, Florida
  - Research Site, North Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Buford, Georgia
  - Research Site, Conyers, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, Noblesville, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Bethesda, Maryland
  - Research Site, High Point, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Friendswood, Texas
  - Research Site, Gonzales, Texas
  - Research Site, Harlingen, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Riverton, Utah
  - Research Site, Alexandria, Virginia
  - Research Site, Portsmouth, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
- United Kingdom (5):
  - Research Site, Bournemouth
  - Research Site, Hayle
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] CDC. (Centers for Disease Control and Prevention). Coronavirus Disease 2019 (COVID-19), Symptoms of Coronavrus. https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html. Published 2020. Accessed 01 July 2020.
- [Background] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Background] Li F. Structure, Function, and Evolution of Coronavirus Spike Proteins. Annu Rev Virol. 2016 Sep 29;3(1):237-261. doi: 10.1146/annurev-virology-110615-042301. Epub 2016 Aug 25. PMID 27578435
- [Background] Miettinen O, Nurminen M. Comparative analysis of two rates. Stat Med. 1985 Apr-Jun;4(2):213-26. doi: 10.1002/sim.4780040211. PMID 4023479
- [Background] WHO. WHO Coronavirus Disease (COVID-19) Dashboard. 2020a.
- [Background] WHO. WHO R&D Blueprint COVID-19 Therapeutic Trial Synopsis Draft 18 February 2020. https://www.who.int/blueprint/priority-diseases/key-action/COVID-19_Treatment_Trial_Design_Master_Protocol_synopsis_Final_18022020.pdf. Published 2020b. Accessed 25 September 2020.
- [Background] Xie Y, Wang Z, Liao H, Marley G, Wu D, Tang W. Epidemiologic, clinical, and laboratory findings of the COVID-19 in the current pandemic: systematic review and meta-analysis. BMC Infect Dis. 2020 Aug 31;20(1):640. doi: 10.1186/s12879-020-05371-2. PMID 32867706
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648
- [Derived] Levin MJ, Ustianowski A, De Wit S, Beavon R, Thissen J, Seegobin S, Dey K, Near KA, Streicher K, Kiazand A, Esser MT. Efficacy, Safety, and Pharmacokinetics of AZD7442 (Tixagevimab/Cilgavimab) for Prevention of Symptomatic COVID-19: 15-Month Final Analysis of the PROVENT and STORM CHASER Trials. Infect Dis Ther. 2024 Jun;13(6):1253-1268. doi: 10.1007/s40121-024-00970-x. Epub 2024 May 4. PMID 38703336
- [Derived] Levin MJ, Ustianowski A, Thomas S, Templeton A, Yuan Y, Seegobin S, Houlihan CF, Menendez-Perez I, Pollett S, Arends RH, Beavon R, Dey K, Garbes P, Kelly EJ, Koh GCKW, Ivanov S, Near KA, Sharbaugh A, Streicher K, Pangalos MN, Esser MT; COVID-19 Study to Optimally Reduce Morbidity in CareHomes and Sites with Enhanced Risk (STORMCHASER) Study Group. AZD7442 (Tixagevimab/Cilgavimab) for Post-Exposure Prophylaxis of Symptomatic Coronavirus Disease 2019. Clin Infect Dis. 2023 Apr 3;76(7):1247-1256. doi: 10.1093/cid/ciac899. PMID 36411267
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00003&attachmentIdentifier=c35deefb-0c9a-4d5c-a910-53a4f500f0e0&fileName=Redacted_Clinical_Study_report_Synopsis.pdf&versionIdentifier=
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00003&attachmentIdentifier=373a042b-d2b9-4e49-b28d-f4c27ee2c31e&fileName=d8850c00003-csp-v6_Redacted.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00003&attachmentIdentifier=f6878577-9ca6-411b-8de2-e4211cd9ffe0&fileName=d8850c00003-sap-v-3-1_redacted_19july_1.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Target sample size was 1125. As this was a multi-site study there was a lag on the information of the number of participants recruited, hence we ended up with a population slightly over 1125 (N=1131).
Groups:
- AZD7442: Single dose 300 mg IM (AZD8895 and AZD1061)
- Placebo: Saline Placebo
Period: Overall Study
Arm/Group | AZD7442 | Placebo
Started | 756 | 375
Dosed (Full Analysis Set) | 749 | 372
Completed | 624 | 304
Not Completed | 132 | 71
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 82 | 38
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 37 | 24
Not completed — Not specified elsewhere | 8 | 6

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7442 | Placebo | Total
Number analyzed (Participants) | 749 | 372 | 1121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.62 (15.74) | 45.97 (16.20) | 46.40 (15.89)
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 48.00 [18 to 92] | 47.00 [18 to 89] | 48.0 [18 to 92]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full Analysis Set
  Participants
    Female | 375 | 182 | 557
    Male | 374 | 190 | 564
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    American Indian or Alaska Native | 6 | 1 | 7
    Asian | 15 | 13 | 28
    Black or African American | 76 | 36 | 112
    Multiple | 4 | 4 | 8
    Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
    Not reported | 15 | 3 | 18
    Unknown | 3 | 0 | 3
    White | 628 | 314 | 942
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    Hispanic or Latino | 435 | 210 | 645
    Not Hispanic or Latino | 299 | 159 | 458
    Not reported | 11 | 1 | 12
    Unknown | 4 | 2 | 6
Any COVID-19 comorbidities at baseline [Count of Participants; unit: Participants]
  Yes | 418 | 210 | 628
  MISSING | 331 | 162 | 493
Any high risk for severe COVID-19 at baseline [Count of Participants; unit: Participants]
  Yes | 486 | 243 | 729
  MISSING | 263 | 129 | 392
SARS-CoV-2 status at baseline [Count of Participants; unit: Participants]
  Negative | 651 | 327 | 978
  Positive | 34 | 14 | 48
  MISSING | 64 | 31 | 95
Baseline BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Data has not been recorded for 3 subjects in the AZD7442 arm
  kg/m^2
    number analyzed (Participants) | 746 | 372 | 1118
    (all) | 29.60 (6.67) | 29.80 (6.68) | 29.67 (6.67)
Height [Mean (Standard Deviation); unit: cm] — Population: Data has not been recorded for 3 subjects in the AZD7442 arm
  cm
    number analyzed (Participants) | 746 | 372 | 1118
    (all) | 168.43 (10.56) | 168.57 (10.32) | 168.5 (10.48)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Case of SARS-CoV-2 RT-PCR Positive Symptomatic Illness
Description: To estimate the efficacy of a single IM dose of AZD7442 compared to placebo for the prevention of COVID-19
Time Frame: Planned to be evaluated through Day 183, however, the number of participants required was achieved 127 days after the study start date
Population: All randomized participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 749 | 372
Participants
  Primary Analysis | 23 | 17
  Final analysis | 28 | 24
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; Test type: Superiority; p = 0.212, Poisson regression; Relative Risk Reduction = 33.31, 95% CI 2-sided [-25.92 to 64.68] — Primary Analysis Estimates are based on Poisson regression with robust variance. The model includes covariate for treatment and the log of follow-up time as an offset. Estimated RRR greater than 0% provides evidence in favor of AZD7442
Statistical Analysis 2: Comparison: AZD7442 vs Placebo; Test type: Superiority; p = 0.044, Poisson regression; Relative Risk Reduction = 43.28, 95% CI 2-sided [1.40 to 67.37] — Final Analysis Estimates are based on Poisson regression with robust variance. The model includes covariate for treatment and the log of follow-up time as an offset. Estimated RRR greater than 0% provides evidence in favor of AZD7442

2. Primary Outcome: AEs, SAEs, MAAEs, and AESIs Post Dose of IMP
Time Frame: 457 Days
Measure: Number; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 749 | 372
Participants
  Any Adverse Event | 348 | 193
  Non-serious Adverse Event | 345 | 191
  Serious Adverse Events | 20 | 16
  Medically Attended Adverse Events | 95 | 52
  Adverse Events of Special Interest | 4 | 4

3. Secondary Outcome: The Incidence of SARS-CoV-2 RT-PCR-positive Severe or Critical Symptomatic Illness Occurring After Dosing With IMP
Time Frame: 183 Days
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 749 | 372
Participants
  Primary analysis | 0 | 1
  Final Analysis | 0 | 1
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; Test type: Superiority; p = 0.664, Poisson regression; Relative Risk Reduction = 100, 97.5% CI 1-sided [lower limit -1836.98]

4. Secondary Outcome: The Incidence of Participants Who Have a Post-treatment Response (Negative at Baseline to Positive at Any Time Post-baseline) for SARSCoV- 2 Nucleocapsid Antibodies
Time Frame: 366 Days
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 570 | 281
Participants | 173 | 98
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; Test type: Superiority; p = 0.163, Poisson regression; Relative Risk Reduction = 13.90, 95% CI 2-sided [-6.23 to 30.21]

5. Secondary Outcome: The Incidence of COVID-19-related Death Occurring After Dosing With IMP
Time Frame: 366 Days
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 749 | 372
Participants | 0 | 0

6. Secondary Outcome: The Incidence of All-cause Mortality Occurring After Dosing With IMP
Time Frame: 366 Days
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 749 | 372
Participants | 3 | 2
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; Test type: Superiority; p = 0.744, Poisson regression; Relative Risk Reduction = 25.75, 95% CI 2-sided [-343.53 to 87.57]

7. Secondary Outcome: Serum AZD7442 Concentrations, PK Parameters
Time Frame: 457 Days
Population: Only AZD7442 arm samples have been analysed for PK concentrations. Baseline and Day 457 were not calculated due to lot of missing samples or concentrations < LLOQ
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 722 | 0
µg/mL
  Day 8: number analyzed (Participants) | 665 | 0
  Day 8 | 10.028 (110.166) |
  Day 29: number analyzed (Participants) | 667 | 0
  Day 29 | 11.718 (72.721) |
  Day 58: number analyzed (Participants) | 641 | 0
  Day 58 | 9.420 (75.160) |
  Day 92: number analyzed (Participants) | 659 | 0
  Day 92 | 7.183 (81.706) |
  Day 183: number analyzed (Participants) | 645 | 0
  Day 183 | 2.975 (79.694) |
  Day 366: number analyzed (Participants) | 585 | 0
  Day 366 | 0.696 (63.725) |

8. Secondary Outcome: Incidence of ADA to AZD7442 in Serum
Time Frame: 457 Days
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 629 | 326
Participants | 110 | 6

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | AZD7442 | Placebo
All-Cause Mortality (participants affected / at risk) | 3/749 | 2/372
Serious Adverse Events (participants affected / at risk) | 20/749 | 16/372
Other Adverse Events (participants affected / at risk) | 345/749 | 191/372
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442 (N=749) | Placebo (N=372)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Bipolar i disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442 (N=749) | Placebo (N=372)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Mycotic allergy (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 2 (2)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Asymptomatic covid-19 (Infections and infestations) | 7 (7) | 5 (5)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 6 (6) | 3 (3)
Covid-19 (Infections and infestations) | 117 (125) | 53 (54)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (4) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 2 (2)
Epstein-barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (2)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 16 (17) | 4 (6)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 4 (4) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 3 (3) | 2 (2)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 7 (7) | 4 (5)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Suspected covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 3 (3)
Urinary tract infection (Infections and infestations) | 22 (24) | 13 (15)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (5)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (7) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 4 (7) | 5 (12)
Alanine aminotransferase abnormal (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (5)
Aspartate aminotransferase abnormal (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 4 (4)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 12 (15) | 4 (4)
Blood creatinine increased (Investigations) | 2 (3) | 1 (1)
Blood glucose increased (Investigations) | 5 (5) | 1 (1)
Blood iron decreased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 3 (3) | 2 (2)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 9 (10) | 3 (3)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 8 (8) | 4 (4)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 2 (2)
Haematocrit decreased (Investigations) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0)
Influenza a virus test positive (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 2 (2) | 0 (0)
Lymph node palpable (Investigations) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Red blood cells urine (Investigations) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 3 (3) | 0 (0)
White blood cells urine positive (Investigations) | 4 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 7 (7)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (29) | 27 (30)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 18 (18) | 14 (14)
Anosmia (Nervous system disorders) | 18 (18) | 13 (13)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0)
Central pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Dizziness exertional (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 86 (109) | 52 (61)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 2 (3)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (2)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 3 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Glycosuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Hyperplasia adrenal (Endocrine disorders) | 1 (1) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 3 (4)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (5) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic congestion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 80 (95) | 46 (58)
Eye movement disorder (Eye disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (33) | 14 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 50 (64) | 34 (41)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 59 (71) | 28 (34)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 61 (73) | 27 (32)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 3 (3)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Cullen's sign (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Behcet's syndrome (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 11 (11) | 5 (5)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Visceral congestion (Vascular disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 19 (22) | 23 (28)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (24) | 23 (26)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 4 (4) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (10) | 7 (7)
Asthenia (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 32 (34) | 23 (26)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Energy increased (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 57 (67) | 39 (50)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 4 (4) | 2 (3)
Injection site pain (General disorders) | 3 (3) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 7 (7) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 39 (44) | 35 (40)
Pyrexia (General disorders) | 46 (57) | 32 (34)
Swelling (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Results are reported for the Primary analysis conducted during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT04625972/Prot_004.pdf
  • Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT04625972/SAP_005.pdf